CLINICAL TRIAL: NCT06658288
Title: Comparative Effects of Rebound Training and Theraband Resistance Exercise on Agility, Power and Dynamic Balance in Badminton Players With Patellofemoral Pain Syndrome
Brief Title: Comparative Effects of Rebound Training and Theraband Resistance Exercise in Badminton Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0413
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy
Keywords: Agility; Dynamic balance; Power; Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Masking Description: The participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 12 Participants will be in experimental group A. They will perform rebound training for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Rebound Training
- Group B (Experimental): 12 Participants will be in experimental group B. They will perform theraband resistance exercise for six weeks. Measure all values before giving them protocol and after protocol.
  Interventions: Other: Theraband resistance exercise

INTERVENTIONS:
Other: Rebound Training — 12 participants will be in experimental group A giving them rebound training.
  Arms: Group A
Other: Theraband resistance exercise — 12 participants will be in experimental group A giving them theraband resistance exercise with different band resistnce.
  Arms: Group B

SUMMARY:
Comparative Effects of Rebound Training and Theraband Resistance Exercise in Badminton Players With Patellofemoral Pain Syndrome

DETAILED DESCRIPTION:
Comparative Effects of Rebound Training and Theraband Resistance Exercise on agility, power and dynamic balance in Badminton Players With Patellofemoral Pain Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18 to 25 years
* Positive Patellofemoral Compression Test ( Pain is in around the patella and back of knee cap) With playing experience of 3 years will be included
* Minimum Sports activity 1 hour 4 times a week

Exclusion Criteria:

* Recreational players
* Players with recent injury in past 6 months
* Any musculoskeletal and neurological problem
* Player addicted to any drug or alcohol will be excluded

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female only
Enrollment: 24 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Numeric Pain Rating Scale NPRS is based on 11-point numerical rating scale for determining pain intensity, 0(no pain) to 10(worst pain imaginable) pain intensity .NRS pain has high validity and reliability (β = 0.42 [95% CI 0.04, 0.80]
Agility T Test | 6 Weeks
  Agility will be measured by the agility T - tests high intra-trail reliability of the test (ICC=0.98). The participants were instructed to run 9.14 meters from the starting line to the first cone, touch the tip with their right hand, shuffle 4.57 meters to the left to the second cone, shuffle 9.14 meters to the right to the third cone, touch with their right hand, shuffle 4.57 meters to the left to the middle cone, touch with their left hand, and then back pedal to the starting line.
Vertical Jump Power Test | 6 Weeks
  To mark the wall at the height of their jump, the participant applies chalk to the tips of their fingers. After standing away from the wall, the individual uses both arms and legs to help project their body upwards and jumps as high as they can. At the peak of the jump, try to make contact with the wall. Power will be measured by Sargent Test. Vertical Jump test is a very common test for measuring explosive leg power intra rater class reliability ICC = 0.903 to 0.934)
40-Yd Speed Test | 6 Weeks
  Speed will be measured by 40-Yd Sprint Test. The test involves running a single maximum sprint over 40 yards, with the time recorded. The aim of this test will be determine 40-Yd Sprint. Sprints of 40 yd were used to determine quickness ICC > 0.987
Star Excursion Dynamic Balance | 6 Weeks
  The SEBT is a functional test that incorporates a single-leg stance on one leg with maximum reach of the opposite leg. The SEBT is performed with the subject standing at the center of a grid placed on the floor, with 8 lines extending at 45° increments from the center of the grid. The 8 lines positioned on the grid are labeled according to the direction of excursion relative to the stance leg. The plane was constructed in a facility with the help of protractor and adhesive tape on the hard tile floor. Dynamic balance check with balance with Star Excursion Balance Test (SEBT) the intra class correlation coefficients ( 0.86 to 0.92)

CONTACTS AND LOCATIONS:
Overall Officials: Noor Fatima, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, Lynch AD, Snyder-Mackler L, McDonough CM. Patellofemoral Pain. J Orthop Sports Phys Ther. 2019 Sep;49(9):CPG1-CPG95. doi: 10.2519/jospt.2019.0302. PMID 31475628
- [Background] Sisk D, Fredericson M. Update of Risk Factors, Diagnosis, and Management of Patellofemoral Pain. Curr Rev Musculoskelet Med. 2019 Dec;12(4):534-541. doi: 10.1007/s12178-019-09593-z. PMID 31773479
- [Background] Lee JH, Jang KM, Kim E, Rhim HC, Kim HD. Static and Dynamic Quadriceps Stretching Exercises in Patients With Patellofemoral Pain: A Randomized Controlled Trial. Sports Health. 2021 Sep-Oct;13(5):482-489. doi: 10.1177/1941738121993777. Epub 2021 Feb 20. PMID 33615901
- [Background] Lee JH, Shin KH, Han SB, Sun Hwang K, Lee SJ, Jang KM. Prospective comparative study between knee alignment-oriented static and dynamic balance exercise in patellofemoral pain syndrome patients with dynamic knee valgus. Medicine (Baltimore). 2022 Sep 16;101(37):e30631. doi: 10.1097/MD.0000000000030631. PMID 36123932
- [Background] Zambarano EK, Bazett-Jones DM, de Oliveira Silva D, Barton CJ, Glaviano NR. Confidence and Knowledge of Athletic Trainers in Managing Patellofemoral Pain. J Athl Train. 2022 Jan 1;57(1):79-91. doi: 10.4085/1062-6050-0279.21. PMID 35040987
- [Background] Emamvirdi M, Letafatkar A, Khaleghi Tazji M. The Effect of Valgus Control Instruction Exercises on Pain, Strength, and Functionality in Active Females With Patellofemoral Pain Syndrome. Sports Health. 2019 May/Jun;11(3):223-237. doi: 10.1177/1941738119837622. Epub 2019 Apr 29. PMID 31034336
- [Background] Saad MC, Vasconcelos RA, Mancinelli LVO, Munno MSB, Liporaci RF, Grossi DB. Is hip strengthening the best treatment option for females with patellofemoral pain? A randomized controlled trial of three different types of exercises. Braz J Phys Ther. 2018 Sep-Oct;22(5):408-416. doi: 10.1016/j.bjpt.2018.03.009. Epub 2018 Apr 4. PMID 29661570
- [Background] Tramontano M, Pagnotta S, Lunghi C, Manzo C, Manzo F, Consolo S, Manzo V. Assessment and Management of Somatic Dysfunctions in Patients With Patellofemoral Pain Syndrome. J Am Osteopath Assoc. 2020 Mar 1;120(3):165-173. doi: 10.7556/jaoa.2020.029. PMID 32091560
- [Background] Pereira PM, Baptista JS, Conceicao F, Duarte J, Ferraz J, Costa JT. Patellofemoral Pain Syndrome Risk Associated with Squats: A Systematic Review. Int J Environ Res Public Health. 2022 Jul 28;19(15):9241. doi: 10.3390/ijerph19159241. PMID 35954598
- [Background] da Silva Boitrago MV, de Mello NN, Barin FR, Junior PL, de Souza Borges JH, Oliveira M. Effects of proprioceptive exercises and strengthening on pain and functionality for patellofemoral pain syndrome in women: A randomized controlled trial. J Clin Orthop Trauma. 2021 Apr 19;18:94-99. doi: 10.1016/j.jcot.2021.04.017. eCollection 2021 Jul. PMID 33996453
- [Background] Ramirez-Campillo R, Alvarez C, Gentil P, Loturco I, Sanchez-Sanchez J, Izquierdo M, Moran J, Nakamura FY, Chaabene H, Granacher U. Sequencing Effects of Plyometric Training Applied Before or After Regular Soccer Training on Measures of Physical Fitness in Young Players. J Strength Cond Res. 2020 Jul;34(7):1959-1966. doi: 10.1519/JSC.0000000000002525. PMID 29570574
- [Background] Deng N, Soh KG, Abdullah B, Huang D, Xiao W, Liu H. Effects of plyometric training on technical skill performance among athletes: A systematic review and meta-analysis. PLoS One. 2023 Jul 17;18(7):e0288340. doi: 10.1371/journal.pone.0288340. eCollection 2023. PMID 37459333
- [Background] Yalfani A, Ahmadi M, Asgarpoor A. The effect of kinetic factors of dynamic knee valgus on patellofemoral pain: A systematic review and meta-analysis. J Bodyw Mov Ther. 2024 Jan;37:246-253. doi: 10.1016/j.jbmt.2023.11.001. Epub 2023 Nov 14. PMID 38432813